CLINICAL TRIAL: NCT07215026
Title: Understanding Non-small Cell Lung Cancer (NSCLC) Patient Characteristics, Treatment Patterns and Outcomes Via Cross-sEctional Physicians suRvey-based Chart Audit
Brief Title: Understanding Non-small Cell Lung Cancer Patient Characteristics, Treatment Patterns and Outcomes
Acronym: UNCOVER
Status: Enrolling by invitation | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D9260R00023
Record Dates: First submitted 2025-10-08; First posted 2025-10-10 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Non-small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a retrospective, cross-sectional, non-interventional, multi-country survey-based chart audit study to evaluate real-world treatment patterns, patient clinical profiles, and clinical outcomes among a NSCLC patients receiving at least 1L SACT (Systemic anticancer therapy)

DETAILED DESCRIPTION:
This is a retrospective, cross-sectional, non-interventional, multi-country survey-based chart audit study to evaluate real-world treatment patterns, patient clinical profiles, and clinical outcomes among aNSCLC patients receiving at least 1L SACT in Argentina, Brazil, Mexico, Australia, India, Taiwan, Malaysia, Hong Kong, and Turkey. All patient-level data, including patient demographic and clinical characteristics, treatment history, and clinical outcomes, will be collected retrospectively from existing patient medical records provided by participating physicians, without interference with treatment decisions. Informed consent from individual patients will not be required, as this study describes the analysis of deidentified patient data.

ELIGIBILITY:
Patient Eligibility Criteria - Inclusion Criteria Diagnosis: Confirmed de novo stage IIIB, IIIC, or IV NSCLC.

Biomarker Status:

Either: EGFR mutation present Or: No actionable gene alterations (AGAs) detected (including EGFR, ALK, ROS1, NTRK, BRAF V600E, RET, MET, KRAS, HER2; patients not tested for these also eligible).

Treatment Start Window: Initiated 1L SACT (systemic anticancer therapy) for advanced NSCLC between the date of first Tagrisso® (osimertinib) approval for NSCLC in their country and 31 December 2024.

Age: 18 years or older at time of 1L SACT initiation.

- Exclusion Criteria Concurrent Malignancies: Patients on active treatment for another primary malignancy at 1L SACT initiation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population for the UNCOVER observational study consists of two main groups: participating physicians and their eligible patients. The protocol lays out robust criteria for both, ensuring relevant, high-quality clinical data across diverse regions.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2025-10-27 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Outcomes of interest are real-world overall survival (rwOS) | 12 month
  Definition of rwOS rwOS is defined as the interval between the index date and the date of death due to any cause.
  *Patients who are alive or for whom vital status is unknown at the time of data collection will be censored at the date the patient is last known to be alive.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, New Delhi, India

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org.
  Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information
URL: https://vivli.org/